CLINICAL TRIAL: NCT02044354
Title: A Study of Patient Preference Between Cabazitaxel and Docetaxel in First-line Chemotherapy for Metastatic Castrate-resistant Prostate Cancer
Brief Title: Patient Preference Between Cabazitaxel and Docetaxel in Metastatic Castrate-resistant Prostate Cancer
Acronym: CABA-DOC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013-004243-22; 2013/2072 (Other: CSET number)
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — Docetaxel; cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Do/Ca (Other): Arm Do/Ca : Taxotere 75mg/m2/3w x 4 cycles, followed by Jevtana 25mg/m2/3w x 4 cycles
  Interventions: Drug: Taxotere; Drug: Jevtana
- Ca/Do (Other): Arm Ca/Do : Jevtana 25mg/m2/3w x 4 cycles, followed by Taxotere 75mg/m2/3w x 4 cycles
  Interventions: Drug: Taxotere; Drug: Jevtana

INTERVENTIONS:
Drug: Taxotere
Drug: Jevtana

SUMMARY:
Taxotere is the current standard first-line chemotherapy for mCRPC and may be used as second-line therapy in good responders in first-line (Taxotere rechallenge). Jevtana has demonstrated a survival benefit versus mitoxantrone in patients progressing during or after Taxotere and is now the standard second-line chemotherapy. Taxotere and Jevtana have different toxicity profiles.

Many patients who are receiving Jevtana for second-line treatment indicate they prefer this agent over Taxotere with regards to the general tolerance (namely peripheral neuropathy, nail changes, asthenia). This was not expected since Jevtana in post-Taxotere setting was associated with more grade 3-4 adverse events such as febrile neutropenia and diarrhea than Taxotere in first-line setting.

The study design of CABA-DOC is similar to that of the PISCES trial which evaluated the patient preference between two standard treatments for first-line metastatic kidney cancer. Despite similar PFS improvements over placebo in phase III trials, results clearly showed that patients preferred pazopanib over sunitinib.

A randomized phase III study is currently comparing the efficacy of Taxotere and Jevtana in first-line setting with overall survival as a primary end-point. Assessing patient preference between Jevtana and Taxotere would contribute to further identify differences between these two taxanes and clarify which one of these two taxanes should be used for second-line chemotherapy and perhaps for first-line chemotherapy in the future.

Assessing patient preference between the two taxanes might be less biased in the first-line setting where patients have no previous experience with a taxane.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated to a social security regimen ;
* Male patients older than 18 years ;
* Histologically confirmed adenocarcinoma of the prostate ;
* Continued androgen deprivation therapy either by LHRH agonists/antagonists or orchidectomy ;
* Serum testosterone <0.50 ng/ml (1.7 nmol/L) ;
* Progressive disease (PSA progression or radiological progression or clinical progression) ;
* ECOG 0-2 ;
* Information delivered to patient and informed consent form signed by the patient or his legal representative ;
* Adequate organ or bone marrow function as evidenced by:

  * Hemoglobin >/= 10 g/dL
  * Absolute neutrophil count >/=1.5 x 109/L,
  * Platelet count >/=100 x 109/L,
  * AST/SGOT and/or ALT/SGPT </=1.5 x ULN;
  * Total bilirubin </=1.5 x ULN,
  * Serum creatinine </=1.5 x ULN. If creatinine 1.0 - 1.5 xULN, creatinine clearance will be calculated according to CKD-EPI formula and patients with creatinine clearance <60 mL/min should be excluded

Exclusion Criteria:

* Patients having received an investigational drug and/or prior surgery, radiation, chemotherapy, or other anti-cancer therapy within 4 weeks prior enrolment in the study, excepted radiotherapy directed to a single bone lesions which is nonacceptable if within 2 weeks ;
* Prior treatment with Taxotere or Jevtana ;
* Pre-existing symptomatic peripheral neuropathy grade > 2 (CTCAE V4) ;
* Uncontrolled cardiac arrhythmias, angina pectoris, and/or hypertension. History of congestive heart failure (NYHA III or IV) or myocardial infarction within last 6 months is also not allowed ;
* History of severe hypersensitivity reaction (grade ≥3) to polysorbate 80 containing drugs ;
* Uncontrolled severe illness or medical condition (including uncontrolled diabetes mellitus), active infection including HIV infection, active Hepatitis B or C infection that would preclude participation in the trial ;
* Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a one week wash-out period is necessary for patients who are already on these treatments) ;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2014-05-22 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Patient preference | Assessed up 21 weeks after randomization
  Patient preference (Taxotere versus Jevtana) assessed by a single question after completion of the second period of chemotherapy.
  Primary outcome measure will be assessed in the intent-to-treat population as defined by all patients having completed the first 4 cycles without progression and having received at least 1 cycle of the second treatment period. Patients having progressed during the first period will discontinue the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Fizazi, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, Val de Marne, France

REFERENCES:
- [Derived] Baciarello G, Delva R, Gravis G, Tazi Y, Beuzeboc P, Gross-Goupil M, Bompas E, Joly F, Greilsamer C, Hon TNT, Barthelemy P, Culine S, Berdah JF, Deblock M, Ratta R, Flechon A, Cheneau C, Maillard A, Martineau G, Borget I, Fizazi K; Groupe d'Etude des Tumeurs Uro-Genitales (GETUG).. Patient Preference Between Cabazitaxel and Docetaxel for First-line Chemotherapy in Metastatic Castration-resistant Prostate Cancer: The CABADOC Trial. Eur Urol. 2022 Mar;81(3):234-240. doi: 10.1016/j.eururo.2021.10.016. Epub 2021 Nov 14. PMID 34789394